CLINICAL TRIAL: NCT02005523
Title: Study of RNS60 on Post-operative Pain and Function in Patients Undergoing Hip Labral Repair or Reconstruction Surgery
Brief Title: Study of RNS60 on Pain and Function After Hip Labral Repair
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Revalesio Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 07.1.1.H2
Record Dates: First submitted 2013-12-03; First posted 2013-12-09 (Estimated); Last update posted 2015-02-06 (Estimated); Status verified 2015-02

CONDITIONS: Hip Labral Tear
MeSH Terms: interventions — RNS60; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- RNS60 (Experimental)
  Interventions: Drug: RNS60
- Saline (Placebo Comparator)
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: RNS60
  Arms: RNS60
Drug: Saline
  Arms: Saline

SUMMARY:
The purpose of this study is to see if use of RNS60 during hip labral repair surgery decreases pain and improves functional capacity post-operation.

Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Assessment of post-operative pain | 1 week
  Comparison of scores from validated pain scales from post-surgery to one week.

CONTACTS AND LOCATIONS:
Locations (1):
- Tacoma, Washington, United States